CLINICAL TRIAL: NCT05683262
Title: Does Combining USG-Guided Coccygeal Nerve Block with Sacrococcygeal And/or Intercoccygeal Joint Injection Have an Additive Effect on the Treatment of Coccydynia? Comparison of Functional Outcomes: a Prospective, Randomized, Double-Blind Study
Brief Title: The Effect of USG-Guided Coccygeal Nerve Block on Sacrococcygeal And/or Intercoccygeal Joint Injection for Coccydynia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aslinur Keles Ercisli, MD, Principal Investigator, Fatih Sultan Mehmet Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E-83041234-604.16.01-8011
Record Dates: First submitted 2022-12-24; First posted 2023-01-13 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Coccyx Disorder; Coccygodynia; Coccyx Injury
Keywords: Coccydynia; Coccygeal nerve; Ultrasonography; Coccyx

STUDY DESIGN:
Intervention Model Description: Randomised, Double Blind Study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound-guided sacrococcygeal and/or intercoccygeal joint injection (Active Comparator): Ultrasound-guided sacrococcygeal and/or intercoccygeal joint injection is applied to patients in this group
  Interventions: Procedure: Ultrasound-guided sacrococcygeal and/or intercoccygeal joint injection
- Ultrasound-guided sacrococcygeal and/or intercoccygeal joint injection with coccygeal nerve block (Active Comparator): Ultrasound-guided coccygeal nerve blockade is done before the application of ultrasound-guided sacrococcygeal and/or intercoccygeal joint injection to patients in this group
  Interventions: Procedure: Ultrasound-guided coccygeal nerve block; Procedure: Ultrasound-guided sacrococcygeal and/or intercoccygeal joint injection after coccygeal nerve block

INTERVENTIONS:
Procedure: Ultrasound-guided sacrococcygeal and/or intercoccygeal joint injection — Ultrasound guidance is used for correct visualization of injection site, and so obtained more successful results. Patients are placed in the prone position with a pillow under the abdomen to flatten the lumbar curvature. Lower extremities should be internally rotated while feet are inverted to help flatten the gluteal region. Injection site is cleaned thrice with povidone iodine %10 solution and covered with sterile drapes. Ultrasonography gel was applied on the probe and the probe was wrapped with a transparent thin sheath and cleaned with povidone iodine. Sterile gel is applied on the skin. The sacrococcygeal ligament, the sacrococcygeal and intercoccygeal joints were visualized. The sacrococcygeal and/or intercoccygeal joints were entered using the in-plane technique with a 23 gauge 6 cm long needle. When it was seen that the needle tip was inside the joint, 3 cc of 2% lidocaine + 1 cc betamethasone solution was injected.
  Arms: Ultrasound-guided sacrococcygeal and/or intercoccygeal joint injection
Procedure: Ultrasound-guided coccygeal nerve block — Patients are placed in the prone position with a pillow under the abdomen. Lower extremities are internally rotated while feet are inverted. Injection site and the probe are cleaned thrice with povidone iodine %10 solution. Sterile gel is applied. The prob was placed on coccygeal cornu and the coccygeal nerve was visualized superomedial to the CC in the subcutaneous tissue layer. Hydrodissection was made by administering 5 ml of 5% dextrose + 1 ml of 2% lidocaine via an in-plane approach with a 23 gauge 6 cm long needle, targeting the short axes of the bilateral coccygeal nerves.
  Arms: Ultrasound-guided sacrococcygeal and/or intercoccygeal joint injection with coccygeal nerve block
Procedure: Ultrasound-guided sacrococcygeal and/or intercoccygeal joint injection after coccygeal nerve block — After the coccygeal nerve block, when the pain with palpation of the coccygeal region was reduced by at least 50%, the sacrococcygeal ligament, sacrococcygeal and intercoccygeal joints were visualized.The sacrococcygeal and/or intercoccygeal joints were entered using the in-plane technique with a 23 gauge 6 cm long needle. When the needle tip was inside the joint, 3 cc of 2% lidocaine + 1 cc betamethasone solution was injected.
  Arms: Ultrasound-guided sacrococcygeal and/or intercoccygeal joint injection with coccygeal nerve block

SUMMARY:
Coccydynia refers to a significant pain, that does not radiate, in and around the coccyx region. This symptom is typically worsen while sitting, especially on hard surfaces, standing up from sitting position and standing for long time. The steroid and anesthetic injection to the sacrococcygeal, intercoccygeal joints and impar ganglions are the most commonly cited second line management option in the literatures for refractor cases. The coccygeal nerve blockade or radiofrequency ablation is also used for coccydynia especially for traumatic cases. The aim of the study is; to evaluate the efficacy of ultrasound-guided sacrococcygeal and/or intercoccygeal joint injection in coccydynia and to investigate whether coccygeal nerve blockade has an additional contribution to this treatment.

DETAILED DESCRIPTION:
Coccydynia refers to a significant pain, that does not radiate, in and around the coccyx region. This symptom is typically worsen while sitting, especially on hard surfaces, standing up from sitting position and standing for a long time. There are several uncertainties with respect to the origin of etiology and the commonest factor for coccydynia is external and internal trauma such as falling, giving birth. Also there are idiopathic cases. The risk of coccydynia progression is higher in the female gender and when obesity is present. The morphology and hypermobility of coccyx are associated with coccydynia and degenerative changes in the intercoccygeal discs have been incriminated to be a cause of pain in 41% of idiopathic and 44% of traumatic coccydynia. The other causes such as infections, tumors such as chordoma, osteoid osteoma or notochordal cell tumors. The antero-posterior (AP) and lateral radiographs are primary imagining modality to rule out these conditions and also to investigate predisposing factors for coccydynia such as bony spicule, retroverted coccyx, subluxation or scoliosis of coccyx. The radiographs are also useful to find out any fracture or dislocation in cause of trauma. Angular mobility evaluation is done by dynamic imaging modalities and still mostly used method is dynamic radiographs which are performed in standing and seated position at the point of maximum pain. Magnetic resonance imaging (MRI) is used for chronic cases to identify most accurate diagnosis and to find exact irritation point and also for ruling out the infections and tumors. A wide range of treatment options have been described till date and conservative therapy such as heat, ice, seat cushions, topical anesthetic and oral/topical non-steroidal anti-inflammatory drugs and intrarectal/intravaginal manual manipulation is successful in %90 of cases. The second line management option for refractor cases is steroid and anesthetic injections however, site of injection is controversial. The sacrococcygeal, intercoccygeal joints and impar ganglions are the most commonly sites for injections cited in the literatures. The success rate of the sacrococcygeal and intercoccygeal joints injections are reported as 60% in most of the studies and the symptoms of nearly one third of the patients relapse within one year. The coccygectomy is an effective modality for these refractory cases but, postoperative complications lead to continue to search conservative treatments options. The innervation of coccyx posteriorly is mostly done by paired of coccygeal nerves and the posterior rami of fourth and fifth sacral nerves which are joining with coccygeal nerves. The coccygeal nerves innervate the coccygeal periosteum, sacrococcygeal joint and the skin over the coccyx. Pain occur at posterior region, after trauma such as falling or long time sitting may be elicited by coccygeal nerves. The coccygeal nerve emerges from the conus medullaris and pierces the posterior sacrococcygeal ligament while it descends in sacral canal. At the level of coccygeal cornu (CC), it is in the the subcutaneous layer and medial to the CC. Therefore coccygeal nerve blockade or radiofrequency ablation is also used for coccydynia especially for traumatic cases. Image guidance such as ultrasound (USG), fluoroscopy, computerized tomography (CT) provide visualization of the needle into the target and improves the accuracy of injections. The use of USG improve the identification of musculoskeletal structures and it spares the patient radiation exposure. It has advantage over the other modalities in that it is cost effective, portable and adapted in multiple disciplines and it has therapeutic safety.

In this study, it is planned to assessed the change of pain severity of the patients who had sacrococcygeal and/or intercoccygeal joint injection with/without coccygeal nerve block in our clinic due to the complaint of coccydynia resistant to conservative treatment methods, by applying the Numeric Rating Scale (NRS). Patients are asked to indicate rates of their pain on the day of presentation during palpation of coccyx, at the first sitting, sitting on soft and hard surface, standing up from sitting position, standing for long time, during defecation, sexual intercourse and menstrual cycle, and also 1 week, 4 weeks, 3 moths and 6 months after the injection for each. Participants are asked to indicate rates of their pain according to NRS during sitting, standing up from sitting position and on palpation of coccyx at the first hour of injection. The pain elicited by injection is also asked after one hour, to determine the effect of coccygeal nerve block which is applied before the sacrococcygeal and/or intercoccygeal joint injection. The second outcome measurement method is assessing the change of pain-free sitting time as a minute before the injection, and one hour, 1 week, 4 weeks, 3 moths and 6 months after the injection.The Oswestry Disability Index for patients with low back pain, Short Form-12 (SF-12) are applied to the participants before the procedure and, at the 1st month, 3rd months and 6 months after the treatment. In these ways, it is planned to evaluate the efficacy of sacrococcygeal and/or intercoccygeal joint injection and also to understand does any additive effect of coccygeal nerve blockade to this treatment approach.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years
2. Patients who have coccygeal pain and have not benefited from conservative treatment
3. Be able to understand enough Turkish to complete the outcome questionnaire
4. Patients whose informed consent was obtained for participation in the study

Exclusion Criteria:

1. Fibromyalgia
2. History of surgery for coccydynia
3. Pregnancy or breastfeeding
4. Inflammatory disease which effect the spine
5. Malignancy
6. Coagulation disorders
7. Infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Change in pain severity of patients from baseline to each checkpoints | From pre-interventional time to post-interventional 1st hour, first week, 4th week, 3rd month, 6th moth
  Pain of the participants will be assessed by one of the most commonly used pain scale "numerical rating scale". It is numeric version of visual analog scale in which a patient selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing "no pain" to '10' representing "pain as bad as you can imagine". Participant is asked to indicate rates of their pain on the day of presentation during palpation of coccyx, at the first sitting, sitting on soft and hard surface, standing up from sitting position, standing for long time, during defecation, sexual intercourse and menstrual cycle, and also 1 week, 4 weeks, 3 moths and 6 months after the injection for each. Participant is also asked to indicate rates of their pain one hour after the injection during sitting, standing up from sitting position and on palpation of coccyx.
Change in pain-free sitting time of patients from baseline to each checkpoints | From pre-interventional time to post-interventional 1st hour, first week, 4th week, 3rd month, 6th moth
  Participant is asked to indicate pain-free sitting time as a minute on the day of presentation, and one hour, 1 week, 4 weeks, 3 moths and 6 months after the injection. Longer duration indicating better result.
Pain according to NRS during injection | 1st hour
  the pain elicited by injection is asked to participants to determine effect of coccygeal nerve block after one hour of injection. The score ranges from 0 to 10, with 0 indicating "No Pain" and 10 "Worst Imaginable Pain

SECONDARY OUTCOMES:
Change the patient reported quality of life assessment from baseline to each checkpoints | From pre-interventional time to post-interventional 4th week, 3rd month, 6th moth
  Defining the change in quality of life scores of patients using Short Form 12 Health Survey (SF-12). The SF-12 is a standardized health related quality of life outcome questionnaire. The questionnaire consists of 12 items questioned weighted and summed to provide physical and mental health scores (PCS and MCS). The two composite scores are computed using the scores on twelve questions that range from 0 to 100, with higher score indicating better health.
Change the patient reported disability from baseline to each checkpoints | From pre-interventional time to post-interventional 4th week, 3rd month, 6th moth
  The Oswestry Disability Index is an effective method of measuring disability in patients with back and leg pain and is well suited to patients who have had persistent severe disability. The questionnaire consists of 10 items with each item having six statements. All scores are summed, then multiplied by two to obtain the index (range 0 to 100) with higher score indicating greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Feyza Unlu Ozkan, Study Director — Fatih Sultan Mehmet Training and Research Hospital
Locations (1):
- Farih Sultan Mehmet Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sencan S, Edipoglu IS, Ulku Demir FG, Yolcu G, Gunduz OH. Are steroids required in the treatment of ganglion impar blockade in chronic coccydynia? a prospective double-blinded clinical trial. Korean J Pain. 2019 Oct 1;32(4):301-306. doi: 10.3344/kjp.2019.32.4.301. PMID 31569923
- [Background] Garg B, Ahuja K. Coccydynia-A comprehensive review on etiology, radiological features and management options. J Clin Orthop Trauma. 2021 Jan;12(1):123-129. doi: 10.1016/j.jcot.2020.09.025. Epub 2020 Sep 24. PMID 33716437
- [Background] Mitra R, Cheung L, Perry P. Efficacy of fluoroscopically guided steroid injections in the management of coccydynia. Pain Physician. 2007 Nov;10(6):775-8. PMID 17987101
- [Background] Datir A, Connell D. CT-guided injection for ganglion impar blockade: a radiological approach to the management of coccydynia. Clin Radiol. 2010 Jan;65(1):21-5. doi: 10.1016/j.crad.2009.08.007. Epub 2009 Oct 24. PMID 20103417
- [Background] Woon JT, Stringer MD. Clinical anatomy of the coccyx: A systematic review. Clin Anat. 2012 Mar;25(2):158-67. doi: 10.1002/ca.21216. Epub 2011 Jul 7. PMID 21739475
- [Background] Chen Y, Huang-Lionnet JHY, Cohen SP. Radiofrequency Ablation in Coccydynia: A Case Series and Comprehensive, Evidence-Based Review. Pain Med. 2017 Jun 1;18(6):1111-1130. doi: 10.1093/pm/pnw268. PMID 28034983
- [Background] Wu WT, Hsu YC, Chang KV, Ozcakar L. Ultrasound Imaging and Ultrasound-Guided Injection of the Coccygeal Nerve for Coccydynia. Am J Phys Med Rehabil. 2022 Jul 1;101(7):e108-e109. doi: 10.1097/PHM.0000000000001987. Epub 2022 Feb 23. No abstract available. PMID 35220319